# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT04102189 |
| Sponsor trial ID: | NN9536-4451 |
| Official title of study: | Effect and safety of semaglutide 2.4 mg once weekly on weight management in adolescents with overweight or obesity |
| Document date* | 16 December 2021 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated. Note: The date in the header of Page 2 is the date of compilation of the documents and not of an update to content.

Semaglutide
Trial ID: NN9536-4451
Clinical Trial Report
Appendix 16.1.9

Date: 10 March 2022
Version: 1.0
Status: Final

## 16.1.9 Documentation of statistical methods

## List of contents

Statistical analysis plan ...... Link

Redacted statistical analysis plan Includes redaction of personal identifiable information only.

VV-CLIN-134203 1.0

VV-TMF-4906149 | 1.1 | NN9536 - 4451

Statistical Analysis Plan Study ID: NN9536-4451


Date: Version: Status: Page:

16 December 2021 | Novo Nordisk 1.0 Final 1 of 24

Statistical Analysis Plan

Protocol title: Effect and safety of semaglutide 2.4 mg once weekly on weight management in adolescents with overweight or obesity

Substance: semaglutide


#### CONFIDENTIAL

Date: Version: Status: Page:

16 December 2021 Novo Nordisk 1.0 Final


# **Table of contents**

| | | | | | Page |
|---|---|---|---|---|---|
| T | able of | f content | s | | 2 |
| Li | ist of a | hbrevia | ions | | 3 |
| | | _ | | | |
| 1 | | | | | |
| | 1.1 | | | | |
| | | 1.1.1 | | | |
| | | | | mary objective | |
| | | | | ondary objectives | |
| | | 1.1.0 | | ploratory objectives | |
| | | 1.1.2 | | marr actional d | |
| | | | | mary estimandondary estimand | |
| | | 1.1.3 | | ondary estimatio | |
| | | 1.1.3 | • | nary endpoint | |
| | | | | nary endpoint | |
| | | | | oportive secondary endpoints | |
| | | | | ploratory endpoints | |
| | | 1.1.4 | | normory enopolitic | |
| | 1.2 | | | alysis plan | |
| 2 | Stati | stical co | siderations | | 9 |
| | 2.1 | | | | |
| | 2.2 | | | n | |
| | 2.3 | | | s | |
| | 2.4 | | • | | |
| | | 2.4.1 | General conside | erations | 10 |
| | | 2.4.2 | Primary endpoin | nt | 11 |
| | | 2.4.3 | Secondary endp | ooints | 15 |
| | | | | nfirmatory secondary endpoint | |
| | | | | pportive secondary endpoints | |
| | | 2.4.4 | | lpoints | |
| | | 2.4.5 | - | | |
| | | | | ogroup analyses | |
| | 2.5 | - | | iods | |
| | | 2.5.1 | | e of the 95 <sup>th</sup> percentile (CDC.gov) | |
| | | 2.5.2 | | SDS (WHO.int) | |
| | | 2.5.3 | | | |
| 3 | Char | nges to tl | e statistical anal | yses planned in the protocol | 23 |
| 4 | Dofo | noncos | | | 24 |

Date: Version: Status:

Page:

16 December 2021 Novo Nordisk 1.0

Final


## List of abbreviations

available but discontinued AD ADA American Diabetes Association

AE adverse event

ALT alanine aminotransferase ANCOVA analysis of covariance

available on randomised treatment AT

BMI body mass index

Centers for Disease Control and Prevention **CDC** 

COA clinical outcome assessment

CI confidence interval

C-SSRS Columbia Suicidality Severity Rating Scale

**ECG** electrocardiogram

**ETD** estimated treatment difference

**FAS** full analysis set

**FPG** fasting plasma glucose HbA<sub>1c</sub> glycated haemoglobin HDL high density lipoprotein

HOMA-B homeostasis model assessment of beta-cell function homeostasis model assessment of insulin resistance HOMA-IR

International Society for Paediatric and Adolescent Diabetes **ISPAD** 

**IWOOL** Impact of Weight on Quality of Life jump to reference multiple imputation J2R-MI LAO-OT last available observation on-treatment

LDL low-density lipoprotein LR logistic regression

missing and discontinued MD

mixed model for repeated measurements **MMRM** 

missing on randomised treatment MT

odds ratio OR

PHQ-9 Patient Health Questionnaire 9

PK pharmacokinetic

PYE patient years of exposure PYO patient years of observation

RD-MI multiple imputation using retrieved subjects

SAE serious adverse event SAP statistical analysis plan safety analysis set SAS subcutaneous s.c. standard deviation SD

T2D type 2 diabetes

**TEAE** treatment-emergent adverse event tipping-point multiple imputation TP-MI **VLDL** very low-density lipoprotein World Health Organisation WHO

VV-TMF-4906149 | 1.1 | NN9536 - 4451

| Statistical Analysis Plan | | Date: | 16 December 2021 Novo Nor | disk |
|---|---|---|---|---|
| Study ID: NN9536-4451 | CONFIDENTIAL | Version: | 1.0 | |
| | CONFIDENTIAL | Status: | Final | |
| | | Page: | 4 of 24 | |

# Version history

This statistical analysis plan (SAP) is based on the updated protocol for trial NN9536-4451 "Effect and safety of semaglutide 2.4 mg once weekly on weight management in adolescents with overweight or obesity", version 2.0 (06 January 2021).

| SAP Version | Date | Change | Rationale |
|-------------|------|----------------|------------------|
| 1.0 | | Not Applicable | Original version |


Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 Version: 1.0 Status: Final 

## 1 Introduction

Changes to the protocol-planned analyses are described in section  $\underline{3}$ .

#### 1.1 Trial information

## 1.1.1 Objectives

## 1.1.1.1 Primary objective

To compare the effect of semaglutide s.c. once-weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity on weight management in adolescents (ages 12 to <18 years) with overweight or obesity.

### 1.1.1.2 Secondary objectives

To compare the effect of semaglutide s.c. once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in adolescents (ages 12 to <18 years) with overweight or obesity on:

- Cardiovascular risk factors
- Glucose metabolism

To compare the safety and tolerability of semaglutide s.c. once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in adolescents with overweight or obesity.

#### 1.1.1.3 Exploratory objectives

To compare the effect of semaglutide s.c. once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in adolescents (ages 12 to <18 years) with overweight or obesity on:

Clinical Outcome Assessments (COAs)

To compare additional safety and tolerability of semaglutide s.c. once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in adolescents with overweight or obesity.

#### 1.1.2 Estimands

#### 1.1.2.1 Primary estimand

The estimand will quantify the average treatment difference of semaglutide relative to semaglutide placebo after 68 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment or initiation of rescue interventions (weight management drugs or bariatric surgery) ("effectiveness"/"treatment policy" estimand). The estimand will cover all effect-related objectives.

The following expansion of the primary estimand will cover the exploratory endpoint "Change in body mass index from baseline (week 0) to week 52 (%)". The estimand will quantify the average SAP 4451-statistical-analysis-plan | 5 of 24 |

Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 Version: 1.0
Status: Final 

treatment effect of semaglutide relative to semaglutide placebo after 52 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment or initiation of rescue interventions.

The following expansion of the primary estimand will cover the exploratory endpoint "Change in body mass index from baseline (week 0) to week 75 (%)". The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 75 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment or initiation of rescue interventions.

## 1.1.2.2 Secondary estimand

The estimand will quantify the average treatment difference of semaglutide relative to semaglutide placebo after 68 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects had they remained on their randomised treatment for the entire planned duration of the trial and not started any rescue intervention (weight management drugs or bariatric surgery) ("efficacy"/"hypothetical" estimand). The estimand will cover the primary objective.

## 1.1.3 Endpoints

## 1.1.3.1 Primary endpoint

| Endpoint title | Time frame | Unit |
|----------------|-----------------------------------|------|
| Change in BMI | From baseline (week 0) to week 68 | % |

## 1.1.3.2 Confirmatory secondary endpoints

| Endpoint title | Time frame | Unit |
|---|---|---|
| Achieving ≥5% reduction of body weight | From baseline (week 0) to week 68 | Count of subject |

## 1.1.3.3 Supportive secondary endpoints

Effect endpoints:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in body weight | From baseline (week 0) to week 68 | kg |
| Change in body weight | From baseline (week 0) to week 68 | % |
| Change in BMI percentage of the 95 <sup>th</sup> percentile on gender and age-specific growth charts (CDC.gov) <sup>1</sup> | From baseline (week 0) to week 68 | % |
| Change in BMI (standard deviation score) (WHO.int) <sup>2</sup> | From baseline (week 0) to week 68 | Score points |
| Change in waist circumference | From baseline (week 0) to week 68 | cm |
| Change in systolic blood pressure | From baseline (week 0) to week 68 | mmHg |
| Change in diastolic blood pressure | From baseline (week 0) to week 68 | mmHg |
| Change in HbA <sub>1c</sub> | From baseline (week 0) to week 68 | % point, mmol/mol |
| Achieving ≥5% reduction of BMI | From baseline (week 0) to week 68 | Count of subject |


Date: Version: Status: Page:

16 December 2021 Novo Nordisk 1.0


Final

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in fasting plasma glucose | From baseline (week 0) to week 68 | mmol/L, mg/dL |
| Change in fasting insulin | From baseline (week 0) to week 68 | pmol/L, mU/L |
| Change in total cholesterol | From baseline (week 0) to week 68 | mmol/L, mg/dL |
| Change in high density lipoprotein (HDL) cholesterol | From baseline (week 0) to week 68 | mmol/L, mg/dL |
| Change in low density lipoprotein (LDL) cholesterol | From baseline (week 0) to week 68 | mmol/L, mg/dL |
| Change in very low density lipoprotein (VLDL) cholesterol | From baseline (week 0) to week 68 | mmol/L, mg/dL |
| Change in triglycerides | From baseline (week 0) to week 68 | mmol/L, mg/dL |

## Safety endpoints:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Treatment-emergent adverse events (TEAEs) | From baseline (week 0) to week 75 | Count of subject |
| Treatment-emergent serious adverse events (SAEs) | From baseline (week 0) to week 75 | Count of subject |
| Change in pulse | From baseline (week 0) to week 68 | bpm |
| Change in amylase | From baseline (week 0) to week 68 | U/L |
| Change in lipase | From baseline (week 0) to week 68 | U/L |
| Change in calcitonin | From baseline (week 0) to week 68 | ng/L |
| Change in ALT | From baseline (week 0) to week 68 | U/L |

#### **Exploratory endpoints** 1.1.3.4

## Effect endpoints:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in BMI | From baseline (week 0) to week 68 | kg/m² |
| Change in HOMA-B | From baseline (week 0) to week 68 | % |
| Change in HOMA-IR | From baseline (week 0) to week 68 | Score |
| Change in IWQOL-Kids physical comfort | From baseline (week 0) to week 68 | Score points |
| Change in IWQOL-Kids body esteem | From baseline (week 0) to week 68 | Score points |
| Change in IWQOL-Kids social life | From baseline (week 0) to week 68 | Score points |
| Change in IWQOL-Kids family-relations | From baseline (week 0) to week 68 | Score points |
| Change in IWQOL-Kids total | From baseline (week 0) to week 68 | Score points |
| Achieving ≥10% reduction of body weight | From baseline (week 0) to week 68 | Count of subject |
| Change in BMI | From baseline (week 0) to week 52 | % |
| Change in BMI | From baseline (week 0) to week 75 | % |

Safety endpoints for adolescents with T2D:


 Date:
 16 December 2021
 Novo Nordisk

 Version:
 1.0

 Status:
 Final

 Page:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemia episodes | From baseline (week 0) to week 75 | Count of subject |
| Treatment-emergent hypoglycaemic episodes according to ADA/ISPAD classification (both the 2014 <sup>3</sup> and the 2018 <sup>4</sup> definition) | From baseline (week 0) to week 75 | Count of subject |
| Treatment-emergent hypoglycaemic episodes according to Novo Nordisk classification | From baseline (week 0) to week 75 | Count of subject |

### Safety assessments:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Occurrence of anti-semaglutide antibodies | From baseline (week 0) to week 68 | Count of subject |
| Occurrence of anti-semaglutide antibodies | From baseline (week 0) to week 75 | Count of subject |
| Change in bone age assessment, x-ray | From baseline (week 0) to week 68 | years |
| Change in electrocardiogram (ECG) | From baseline (week 0) to week 68 | Count of subject |
| Change in laboratory parameters | From baseline (week 0) to week 68 | |
| Change in pubertal status (Tanner staging) | From baseline (week 0) to week 68 | Count of subject |
| Change in height (standard deviation score) (WHO.int) | From baseline (week 0) to week 68 | Score points |
| Change in mental health assessed by Columbia Suicidality Severity Rating Scale (C-SSRS) | From baseline (week 0) to week 68 | Score points |
| Change in Patient Reported Health Questionnaire 9 (PHQ-9) | From baseline (week 0) to week 68 | Score points |
| Change in ophthalmological evaluation (for subjects with T2D) | From baseline (week 0) to week 68 | Count of subject |

## Pharmacokinetic analysis

The pharmacokinetic analysis will be done as mentioned in the protocol section 10.4.

## 1.1.4 Type of trial

This is a 68-week, randomised, two-arm, double-blinded, multi-centre clinical trial comparing semaglutide s.c. 2.4 mg once-weekly with semaglutide placebo in adolescents with overweight or obesity.

The trial design is provided in the protocol, section 5.

## 1.2 Scope of the statistical analysis plan

This statistical analysis plan (SAP) is based on the updated protocol for trial NN9536-4451 "Effect and safety of semaglutide 2.4 mg once weekly on weight management in adolescents with overweight or obesity", version 2.0 (06 January 2021) and includes more detailed procedures for executing the statistical analyses.

of 24


Date: Version: Status: Page: 16 December 2021 | Novo Nordisk 1.0 Final 9 of 24

## 2 Statistical considerations

## 2.1 Statistical hypotheses

The tests of superiority of s.c. semaglutide 2.4 mg to semaglutide placebo for the primary and confirmatory secondary endpoints are performed using a fixed-sequence statistical strategy.

This strategy tests the endpoints using a predefined hierarchical order; first the primary endpoint change in BMI (%) from baseline (week 0) to week 68 is tested at a significance level of 5%. If superiority of s.c. semaglutide 2.4 mg to semaglutide placebo is not confirmed, then the testing will stop. If superiority is confirmed (two-sided p-value <5%), the test of the confirmatory secondary endpoint subjects achieving ≥5% reduction of body weight will be performed.

## 2.2 Sample size determination

The trial is designed with an effective power of 90% and 72% to detect differences on the primary endpoint and confirmatory secondary endpoint, respectively. The effective power was calculated under the assumption of independence of endpoints by multiplying the respective marginal powers successively which is a conservative approach.

The assumptions for these calculations are conservatively based on findings from the s.c. semaglutide 0.1 mg and 0.2 mg once daily arms in trial NN9536-4153 and are presented in <u>Table 1</u>.

In the analysis approach addressing the primary estimand, week 68 assessments from retrieved subjects are included. These data are also used to impute missing measurements at week 68 for non-retrieved subjects. The imputation is done separately within each treatment arm. However, for the sample size calculations, missing values regardless of treatment arm are assumed to be similar to semaglutide placebo subjects. These assumptions are likely conservative with respect to the power and correspond to the jump to reference sensitivity analysis described below.

Table 1 Assumptions, marginal power and effective power for each endpoint in the hierarchical testing procedure given an anticipated number of 192 randomised subjects

| Order | Endpoint | Assumed mean (±SD) or proportion for completers | | Expected*<br>mean (±SD) or | Expected*<br>difference or | Marginal<br>power | Effective power |
|---|---|---|---|---|---|---|---|
| | | Semaglutide 2.4<br>mg | Semaglutide<br>placebo | proportion | proportion<br>ratio | (%) | (%) |
| 1 | Change in<br>BMI (%) | 10.5 (±10) | 3 (±10) | 8.5 (±11) | 5.5%-points | 90 | 90 |
| 2 | 5% BW<br>responders | 71% | 42% | 63% | 1.5 | 80 | 72 |

<sup>\*</sup>Accounting for reduced treatment effect among non-completers

All above outlined sample size and power considerations are for the primary estimand for the primary endpoint or the confirmatory secondary endpoints (treatment policy strategy). It is assumed that up to 35% of subjects discontinue permanently and 50% of these are retrieved at week 68. Any superiority conclusions will be based on the primary estimand.


Further assumptions for the sample size calculations are that the significance level is 5%, and that subjects are randomised in a 2:1 ratio to semaglutide or semaglutide placebo. The power calculations for continuous endpoints are based on a t-test on the mean difference assuming equal variances whereas for the categorical endpoint it is based on the Pearson chi-square test for two independent proportions.

All subjects in the semaglutide placebo arm are assumed to have same effect as subjects who complete the trial on semaglutide placebo. Retrieved subjects in the semaglutide arm are assumed to have an effect corresponding to half the treatment difference (compared to semaglutide placebo) of subjects who complete the trial on semaglutide. In the semaglutide arm, non-retrieved subjects and subjects with data missing on randomised treatment are assumed to have an effect corresponding to the semaglutide placebo arm.

#### 2.3 Definition of analysis sets

Two analysis sets are defined:

The *full analysis set (FAS)* includes all randomised subjects according to the intention-to-treat principle.

The *safety analysis set (SAS)* includes all randomised subjects exposed to at least one dose of randomised treatment.

Any observation excluded from the analysis database will be documented before database lock with the reason for exclusion provided.

Two observation periods are defined for each subject:

- In-trial: The *in-trial period* is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site
- On-treatment (with trial product): A time-point is considered as 'on-treatment' if any dose of trial product has been administered within the prior 2 weeks (14 days). The *on-treatment period* is defined as all times which are considered on-treatment
  - In general, the on-treatment period will therefore be from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least two consecutive missed doses
  - For the evaluation of AEs and hypoglycaemic episodes the lag time for each on-treatment time interval is 7 weeks (49 days)

The in-trial and on-treatment periods define the patient years of observation (PYO) and patient years of exposure (PYE), respectively, as the total time duration in the periods.

#### 2.4 Statistical analyses

#### 2.4.1 General considerations

The last available and eligible observation at or before randomisation is used as the baseline value. If no assessments are available, the mean value at randomisation across all subjects is used as the baseline value.

Status:

Final


## 2.4.2 Primary endpoint

Definition of primary endpoint % change in BMI.

Change from baseline to week 68 in BMI (%) is defined as:

% change in BMI= 
$$\frac{\text{(BMI at week 68 - BMI at baseline)}}{\text{BMI at baseline}} \times 100$$

## Analyses addressing the primary estimand

The following statistical analyses and imputation methods are designed to address the primary estimand, i.e. to assess the effectiveness of semaglutide 2.4 mg.

The analysis model for % change in BMI is a linear regression (ANCOVA) of % change in BMI on randomised treatment and stratification group (gender \*Tanner stage group) as factors, and baseline BMI (kg/m²) as covariate. The estimated treatment difference between s.c. semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% CI and corresponding p-value.

The superiority tests of semaglutide 2.4 mg vs. semaglutide placebo will be carried out as follows.

Let  $\mu_{\text{semaglutide}}$  and  $\mu_{\text{semaglutide placebo}}$  denote the true mean of % change in BMI for s.c. semaglutide 2.4 mg and semaglutide placebo group, respectively. The null and alternative hypotheses tested are

H: 
$$\mu_{semaglutide} \ge \mu_{semaglutide \ placebo} \ vs$$
  
 $H_A$ :  $\mu_{semaglutide} < \mu_{semaglutide \ placebo}$ .

The hypothesis will be rejected and superiority claimed, if the upper limit of the estimated two-sided 95% CI is below 0.

## Taxonomy of week 68 assessments being available or missing

For each subject a given assessment at week 68 may be available or missing and <u>Table 2</u> describes the taxonomy for this. Note, this is done per assessment not per subject; subjects may be a different type for different assessments (a subject may have "available on treatment (AT)" for weight but "missing on treatment (MT)" for waist circumference).

Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 | Novo Nordisk
Version: 1.0
Status: Final

Page:


Table 2 Taxonomy for subjects based on week 68 assessments being available or missing

| Assessment<br>at week 68 | On<br>randomised<br>treatment<br>at week 68 | Type description | Type<br>Abbreviation |
|---|---|---|---|
| Available | Yes | Available on randomised treatment: Subjects who complete the trial on randomised treatment with an assessment at week 68: Includes those that stop and restart trial product. | AT |
| | No | Available but discontinued Subjects who discontinued randomised treatment prematurely but returned to have an assessment at week 68. These are also called retrieved subjects | AD |
| Missing | Yes | Missing on randomised treatment: Subjects who complete the trial on randomised treatment without an assessment at week 68: Includes those that stop and restart trial product. | MT |
| | No | Missing and discontinued: Subjects who discontinued randomised treatment prematurely and did not return to have an assessment at week 68. These are also called non-retrieved subjects | MD |

Handling of missing week 68 values for the primary estimand

All available data at week 68 (AT and AD) are used and missing values (MT and MD) at week 68 will be imputed. Several approaches for imputation will be applied. First, a description of the primary imputation approach to address the primary estimand for the primary endpoints is given followed by a description of the sensitivity analyses used to assess the robustness of the primary analysis results. The sensitivity analyses investigate how assumptions on BMI development after discontinuation of randomised treatment impact the estimated treatment contrasts between s.c. semaglutide 2.4 mg and semaglutide placebo. An illustration of all imputation approaches for the primary estimand is given in Figure 1.

Date:

Version:

Status: Page:



Figure 1 Illustration of imputation approaches for the effectiveness estimand Primary imputation approach for the primary estimand

Multiple imputation approach using retrieved subjects (RD-MI): The primary imputation approach for the primary estimand is a multiple imputation similar to the one described by McEvoy<sup>2</sup>.

Missing BMI measurements at week 68 for non-retrieved subjects (MD) are imputed using assessments from retrieved subjects (AD) in each randomised treatment arm. This will be done according to the timing of last available observation during the on-treatment period (LAO-OT) of BMI. Missing BMI measurements at week 68 for subjects on randomised treatment (MT) are imputed by sampling from available measurements at week 68 from subjects on randomised treatment (AT) in the relevant randomised treatment arm. The multiple imputation approach is done in three steps:

1. **Imputation**: Defines an imputation model using retrieved subjects (AD) from FAS and done within groups defined by randomised treatment. The model will be a linear regression of BMI (kg/m<sup>2</sup>) at week 68 on stratification group (gender\*Tanner stage group) as a factor and baseline BMI (kg/m<sup>2</sup>), timing of LAO-OT of BMI (kg/m<sup>2</sup>) and LAO-OT of BMI (kg/m<sup>2</sup>) as covariates. No interactions will be included. If any subjects are MT, an imputation model for missing BMI measurements at week 68 for MT subjects will also be defined using AT subjects in a similar way. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 BMI values for each randomised treatment arm. This will be done 1000 times and result in 1000 complete data sets


Page:


- 2. **Analysis**: Analysis of each of the 1000 complete data sets, using the analysis model (ANCOVA), resulting in 1000 estimations
- 3. **Pooling**: Integrate the 1000 estimation results into a final result using Rubin's formula

Based on NN9536-4153 phase 2 results 1,000 copies should be sufficient to establish stable results. If 1,000 copies are insufficient, 10,000 copies will be used. The multiple imputations will be generated using Novo Nordisk trial number 95364451 as seed number.

Sensitivity analyses

Jump to reference multiple imputation approach (J2R-MI): Missing values of BMI at week 68 (MT and MD) for both the semaglutide 2.4 mg and semaglutide placebo group is by sampling among all available assessments at week 68 in the semaglutide placebo group (AT and AD). This approach makes the assumption that subjects instantly after discontinuation lose any effect of randomised treatment beyond what can be expected from semaglutide placebo treatment as adjunct to diet and physical activity<sup>5</sup>. The multiple imputation approach is done as above with the first step replaced by:

1. Imputation: Defines an imputation model using semaglutide placebo subjects from FAS with a week 68 measurement (AT and AD). The model will be a linear regression of BMI (kg/m²) at week 68 on stratification group (gender\*Tanner stage group) as a factor and baseline BMI (kg/m²) as covariate. No interactions will be included. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 BMI values for each randomised treatment arms. This will be done 1000 times and result in 1000 complete data sets.

The jump to reference approach is the basis for the sample size calculations.

Tipping-point multiple imputation analysis (TP-MI): This analysis will be performed only if superiority is concluded with respect to the primary endpoint. First, missing data are imputed according to the primary multiple imputation approach. Then, a penalty is added to the imputed values at week 68. The approach is to explore a range of penalties for both treatment groups, and the impact these would have on the study conclusions. The 2-dimensional space of penalties covering the range from -30% to 30% will be explored for both treatment groups. This sensitivity analysis evaluates the robustness of the superiority conclusions to departures from the observed change in body weight in both treatment groups.

Excluding subjects from site : In Belgium site where six subjects were randomised it was discovered after all six subjects had been randomised that the stadiometer was not calibrated. A sensitivity analysis of the primary endpoint will be performed in which these six subjects are excluded.

Mixed model for repeated measurements (MMRM): This 'MMRM for effectiveness' will use all assessments regardless of adherence to randomised treatment, including assessments at week 68 for retrieved drop-outs (AD). The MMRM for effectiveness will be fitted using the same factor and covariate as for the primary analyses all nested within visit. An unstructured covariance matrix for

Page:

measurements within the same subject will be employed, assuming that measurements for different subjects are independent.

ANCOVA assuming unequal variances: An alternative analysis model similar to the primary analysis model (ANCOVA), following the primary imputation approach (RD-MI), but assuming unequal variances instead of equal variances. The analysis model for % change in BMI is a linear regression (ANCOVA) of % change in BMI on randomised treatment and stratification group (gender \*Tanner stage group) as factors, and baseline BMI (kg/m<sup>2</sup>) as covariate. The estimated treatment difference between s.c. semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% CI and corresponding p-value.

## Analysis addressing the secondary estimand

The secondary estimand for % change in BMI addresses the efficacy of semaglutide 2.4 mg and will be assessed using a 'MMRM for efficacy'. Week 68 assessments for retrieved subjects (AD) are not used in this analysis. The MMRM for efficacy will use assessments only from subjects who are taking the randomised treatment until end of trial or at first discontinuation of randomised treatment. The derived date of the second consecutive missed dose will be used as the latest date for assessments included in this MMRM. The assessment closest in time and before the derived date of the second consecutive missed dose will be used as last assessment on randomised treatment. For subjects who initiate rescue interventions (weight management drugs or bariatric surgery) before completion or first discontinuation of randomised treatment, the date of starting weight management drugs or undergoing bariatric surgery will be used as last assessment on randomised treatment. The MMRM for efficacy will be fitted using % change in BMI and the same factor and covariate as for the primary analysis all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent.

#### 2.4.3 Secondary endpoints

#### 2.4.3.1 Confirmatory secondary endpoint

The confirmatory secondary endpoint is weight loss ≥5% at week 68 (Yes/No) (≥5% body weight responder endpoint), and is included in the fixed-sequence statistical strategy described above.

## Analysis addressing the primary estimand

The  $\geq$ 5% body weight responder endpoint will be analysed using the same imputation approach as used for the primary endpoint and to address the primary estimand. The imputation model is the same as for the primary endpoint, with BMI replaced by body weight, and the resulting imputed values will then be dichotomized to derive the responder endpoint. The statistical model for the ≥5% body weight responder endpoint is a logistic regression using randomised treatment and stratification group (gender \*Tanner stage group) as factors, and baseline body weight (kg) as a covariate. The estimated odds ratio (OR) between semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% CI and corresponding p-value.

The superiority tests of semaglutide 2.4 mg vs. semaglutide placebo will be carried out as follows for the two analysis models.

Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 Version: 1.0
Status: Final 

Let OR<sub>semaglutide/placebo</sub> denote the true odds ratio between semaglutide 2.4 mg and semaglutide placebo. The null and alternative hypotheses tested are

H: 
$$OR_{\underbrace{semaglutide}_{placebo}} \le 1 \text{ vs}$$
  
 $H_A$ :  $OR_{\underbrace{semaglutide}_{placebo}} > 1$ .

The hypothesis will be rejected and superiority claimed, if the lower limit of the estimated two-sided 95% CI is above 1.

Sensitivity analysis for the confirmatory secondary endpoint: A sensitivity analysis considering non-retrieved subjects as non-responders will be carried out.

## Analyses addressing the secondary estimand

The secondary estimand for the  $\geq$ 5% body weight responder endpoint will be assessed using the same MMRM as for the primary endpoint. Subjects who are missing week 68 body weight will be replaced by predicted values for % weight change at week 68 from the MMRM, and these predicted values will then be dichotomized to derive the responder endpoint. A logistic regression model with randomised treatment as a factor and baseline body weight (kg) as a covariate will then be used to analyse the 5% responder endpoint.

For all analyses of responder endpoints ( $\geq$ 5% body weight reduction,  $\geq$ 10% body weight reduction, and  $\geq$ 5% BMI reduction), in addition to the estimated OR, the estimated treatment differences (ETDs) will be provided by calculating the responder probabilities and treatment differences between responder probabilities based on the logistic regression model, with confidence intervals for treatment differences obtained using the delta method.

An overview of all analysis and imputation methods to address the effectiveness and efficacy estimands for the primary and confirmatory secondary endpoint is given in <u>Table 3</u>.

Table 3 Analysis and imputation methods to address the effectiveness and efficacy estimands for the primary and confirmatory secondary endpoints in the statistical testing hierarchy

| Objective | Endpoint | Test<br>order | Endpoint<br>type | Estimand | Analysis<br>set | Statistical<br>model | Imputation approach | Sensitivity<br>analyses |
|---|---|---|---|---|---|---|---|---|
| Primary er | ıdpoint | | | | | | | |
| Primary | % change in BMI | 1 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI<br>TP-MI<br>Excl. MMRM<br>Unequal<br>variance |
| | | | | Secondary | FAS | MMRM | - | - |
| Confirmat | ory secondary endpoir | ıt | | | · | | | |
| Primary | ≥5% body weight responders | 2 | Binary | Primary | FAS | LR | RD-MI | Non-<br>responders |
| | | | | Secondary | FAS | LR | MMRM | - |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; J2R-MI = jump to reference multiple imputation; TP-MI = tipping point multiple imputation; Excl. = sensitivity analysis excluding site ; MMRM = mixed model for repeated measurements; LR = logistic regression.

Test order refers to the order of the endpoint in the statistical test hierarchy outlined in Table 1.

Page:


## 2.4.3.2 Supportive secondary endpoints

Supportive secondary endpoints are listed in section 1.1.3.3.

## Analyses addressing the primary estimand

The effect-related supportive secondary endpoints will be analysed using the same imputation approach as used for the primary endpoint and to address the primary estimand. The imputation model is the same as for the primary endpoint with BMI replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % change in BMI with baseline BMI replaced by the baseline assessment of the endpoint to be analysed.

The statistical model for the responder endpoint relating to BMI will be logistic regression with randomised treatment as a factor and the baseline assessment of the endpoint to be analysed as covariate.

For fasting insulin, lipids and ALT, a multiplicative model will be used, i.e. the ratio between post randomisation measurements and baseline will be calculated instead of differences, and both the dependent variable and covariate will be log-transformed.

## Analyses addressing the secondary estimand

The supportive secondary endpoints which relate to the primary objective will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoint.

## Analysis of safety endpoints

The safety endpoints pulse and ALT will be analysed using an MMRM for efficacy as described in section 1.1.3.2. These analyses will be based on the safety analysis set. For amylase, lipase and calcitonin descriptive statistics will be provided. The analysis of calcitonin will be stratified by gender.

AEs will be defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the ontreatment period (see definition in section 2.3). TEAEs and SAEs will be summarised by descriptive statistics, such as frequencies and rates. No formal statistical inference will be carried out based on the number of TEAEs and SAEs. AEs in the run-in period (prior to randomisation) will be presented in listings.

An overview of all analysis and imputation methods to address the effectiveness and efficacy estimands for supportive secondary endpoints is given in <u>Table 4</u>.


Date: Version: Status: Page: 16 December 2021 Novo Nordisk

1.0 Final 18 of 24

Table 4 Analysis and imputation methods to address the effectiveness and efficacy estimands for supportive secondary endpoints

| Objective | Endpoint | Endpoint | Estimand | Analysis | Statistical | Imputation |
|---|---|---|---|---|---|---|
| <u> </u> | | type | | set | model | approach |
| | secondary endpoints (effect related | | ъ. | LEAG | 13100111 | DD 14 |
| Primary | Weight change (kg) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| | | | Secondary | FAS | MMRM | - |
| Primary | Weight change (%) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| | | | Secondary | FAS | MMRM | - |
| Primary | BMI percentage of the 95 <sup>th</sup> | Continuous | Primary | FAS | ANCOVA | RD-MI |
| | percentile on gender and age-<br>specific growth charts change<br>(CDC.gov) | | Secondary | FAS | MMRM | - |
| Primary | BMI (standard deviation score) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| - | (WHO.int) change | | Secondary | FAS | MMRM | - |
| Primary | Waist circumference change (cm) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| - | | | Secondary | FAS | MMRM | - |
| Primary | Achieving ≥5% reduction of BMI | Binary | Primary | FAS | LR | RD-MI |
| | | | Secondary | FAS | LR | MMRM |
| Secondary | Systolic blood pressure change (mmHg) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | Diastolic blood pressure change (mmHg) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | HbA <sub>1c</sub> change (%, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | FPG change (mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | Fasting insulin change (pmol/L, mIU/L) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | Total cholesterol change<br>(mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | HDL change (mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | LDL change (mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | VLDL change (mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | Triglycerides change (mmol/L, mg/dL) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Supportive | secondary endpoints (safety relate | d) | | | | |
| Secondary | Number of TEAEs | Continuous | - | SAS | - | - |
| Secondary | Number of SAEs | Continuous | - | SAS | - | - |
| Secondary | Pulse change (bpm) | Continuous | - | SAS | MMRM | - |
| Secondary | Amylase change (U/L) | Continuous | - | SAS | Descriptive statistics | - |
| Secondary | Lipase change (U/L) | Continuous | - | SAS | Descriptive statistics | - |
| Secondary | Calcitonin change (ng/L) | Continuous | - | SAS | Descriptive statistics | - |
| Secondary | ALT change (U/L) | Continuous | | SAS | MMRM | |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; MMRM = mixed model for repeated measurements; BMI = body mass index; HbA1c = Hemoglobin A1c; TEAEs = treatment-emergent adverse events; SAEs = serious adverse events.

## 2.4.4 Exploratory endpoints

Exploratory endpoints are listed in section 1.1.3.4.

## Analyses addressing the primary estimand

The effect-related exploratory endpoints will be analysed using the same imputation approach as used for the primary endpoint and to address the primary estimand. The imputation model is the

Status:

Final 19 of 24

same as for the primary endpoint with BMI replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % change in BMI with baseline BMI replaced by the baseline assessment of the endpoint to be analysed.

The statistical model for responder endpoints relating to body weight will be logistic regression with randomised treatment as a factor and the baseline assessment of the endpoint to be analysed as covariate.

For HOMA-B and HOMA-IR, a multiplicative model will be used, i.e. the ratio between post randomisation measurements and baseline will be calculated instead of differences, and both the dependent variable and covariate will be log-transformed.

## Analyses addressing the secondary estimand

The exploratory endpoints measured at week 68 which relate to the primary objective will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoint.

An overview of all analysis and imputation methods to address the effectiveness and efficacy estimands for effect-related exploratory endpoints is given in <u>Table 5</u>.

### Analysis of safety endpoints

Observed data for exploratory safety endpoints and other safety assessments will be summarised by descriptive statistics.

Hypoglycaemic episodes will be summarised by descriptive statistics, such as frequencies and rates. No formal statistical inference will be carried out based on the number of hypoglycaemic episodes.


 Date:
 16 December 2021
 Novo Nordisk

 Version:
 1.0

 Status:
 Final

 Page:

Table 5 Analysis and imputation methods to address the effectiveness and efficacy estimands for exploratory endpoints

| Objective | Endpoint | Endpoint<br>type | Estimand | Analysis set | Statistical<br>model | Imputation approach |
|---|---|---|---|---|---|---|
| Exploratory endpoints (effect related) | | | | | | |
| Primary | BMI change (kg/m <sup>2</sup> ) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| | | | Secondary | FAS | MMRM | - |
| Primary | Achieving ≥10% reduction of | Binary | Primary | FAS | LR | RD-MI |
| | body weight | | Secondary | FAS | LR | MMRM |
| Primary | BMI change to week 52 (%) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Primary | BMI change to week 75 (%) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | HOMA-B change (%) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | HOMA-IR change (score) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | IWQOL-Kids physical comfort | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | change (score) IWQOL-Kids body esteem change (score) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | IWQOL-Kids social life change (score) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | IWQOL-Kids family-relations change (score) | Continuous | Primary | FAS | ANCOVA | RD-MI |
| Secondary | IWQoL-Kids total change (score) | Continuous | Primary | FAS | ANCOVA | RD-MI |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; MMRM = mixed model for repeated measurements; BMI = body mass index; FPG = fasting plasma glucose; HDL = high density lipoprotein; LDL = low density lipoprotein; VLDL = very low density lipoprotein; LR = logistic regression; IWQoL-Kids = Impact of Weight on Quality of Life-Kids for Clinical Trials; PCD = physical comfort domain; BED = body esteem domain; SLD = social life domain; FRD = family relations domain.

## 2.4.5 Other analyses

All collected data that were not defined as endpoints will be summarised by descriptive statistics.

## 2.4.5.1 Subgroup analyses

Subgroup analyses of the primary and the confirmatory secondary endpoint will be carried out addressing both the primary and the secondary estimand using the same imputation approaches and statistical models as used in the analyses of the primary and confirmatory secondary endpoints. The subgroups are defined in <u>Table 6</u>. The results of the subgroup analyses will be presented with treatment contrasts and treatment-by-subgroup interaction p-values in table form and forest plots.

If a treatment arm has less than 5 subjects within a subgroup, the subgroup will be merged with another, until the criteria of at least 5 subjects per treatment arm and subgroup is reached. For ordered subgroups (e.g. age, baseline BMI), the merging will be done according to the order. For unordered subgroups (e.g. race, region), it will be done by merging the subgroups with the lowest number of subjects.

The results of the subgroup analyses will be submitted to authorities and will not be reported in the clinical trial report.

Table 6 Definition of subgroups

| Subgroup | Levels |
|----------|--------------------------------|
| Age | 12 - <15 years; 15 - <18 years |


Date: Version: Status: Page:

16 December 2021 | Novo Nordisk 1.0 Final


| Subgroup | Levels |
|---|---|
| Sex | Female; Male |
| Ethnicity | Hispanic or Latino; Not Hispanic or Latino |
| Race | White; Other |
| Tanner stage | 2-3; 4-5 |
| BMI | <35 kg/m²; 35 - <40 kg/m²; ≥40 kg/m² |
| Region | Europe (Austria, Belgium, Croatia, Ireland, Russian Federation, United Kingdom);<br>North America (USA);<br>South America (Mexico) |
| Region 2 | USA; Non-USA |

## 2.5 Endpoint derivation methods

## 2.5.1 BMI percentage of the 95<sup>th</sup> percentile (CDC.gov)

The growth charts from the CDC consist of a series of percentile curves that illustrate the distribution of selected body measurements in children from Unites States.

The BMI-for-age reference data applies to children and adolescents (2-20 years).

In practice when using the growth reference data, then the age in months is used to look up the 95<sup>th</sup> percentile. E.g. if a subject is 180.2 months when being measured, then the 95<sup>th</sup> percentile to be used is obtained from the 180.5 month reference, since this reference covers the interval from 180 to 180.99 months. According to CDC<sup>1</sup> at a finer age can be obtained using linear interpolation.

Hence, in order to calculate an exact percentage above the 95<sup>th</sup> percentile for a given age in months, linear interpolation of the 95<sup>th</sup> percentile is applied between the lower 95<sup>th</sup> percentile in months and the upper 95<sup>th</sup> percentile in months.

## 2.5.2 BMI and height SDS (WHO.int)

The BMI standard deviation scores (SDS) and the height SDS scores will be calculated using growth reference data for children and adolescents (5-19 years) from WHO<sup>2</sup>. The SDS scores are sometimes referred to as z-scores also.

The z-score for a subject with a BMI y at age t is given as:

$$z = \frac{\left(\left(\frac{y}{M(t)}\right)^{L(t)} - 1\right)}{S(t)L(t)} \qquad if |z| \le 3$$

where L, M and S depend on sex and age in months and can be looked up in the reference data. If the z-score is between -3 and 3 then no adjustment is needed. If the z-score is > 3 then the score is adjusted as follows:

$$z = 3 + \left(\frac{y - SD3pos}{SD23pos}\right) \qquad if \ z > 3$$

where *SD3pos* is the cut-off 3 SD calculated at t by the LMS method<sup>2</sup>:

$$SD3pos = M(t) * (1 + L(t) * S(t) * (3))^{1/L(t)}$$

and *SD23pos* is the difference between the cut-offs 3 SD and 2 SD calculated at *t* by the LMS method:

$$SD23pos = M(t) * (1 + L(t) * S(t) * (3))^{1/L(t)} - M(t) * (1 + L(t) * S(t) * (2))^{1/L(t)}$$

If the z-score is  $\leq$  3 then the score is adjusted as follows:

$$z = -3 + \left(\frac{y - SD3neg}{SD23neg}\right) \qquad if \ z < -3$$

where *SD3neg* is the cut-off -3 SD calculated at *t*, and *SD23neg* is the difference between the cut-offs -2 SD and -3 SD, both calculated by the LMS method:

$$SD3neg = M(t) * (1 + L(t) * S(t) * (-3))^{1/L(t)}$$

$$SD23neg = M(t) * (1 + L(t) * S(t) * (-2))^{1/L(t)} - M(t) * (1 + L(t) * S(t) * (-3))^{1/L(t)}$$

In practice when using the growth reference data, then the age in whole months is used to look up the L, M and S values. E.g. if a subject is 180.2 months when being measured, then the values of L, M and S to use are done for 180 months, i.e. the age is rounded down to the nearest month.

In order use the same derivation with respect to calculating an exact z-score for a given age in months as for the CDC derivations in section 2.5.1, linear interpolation of the z-score is applied between the lower z-score in months and the upper z-score in months.

The height SDS scores are calculated in the same manner as for the BMI SDS scores.

Some subjects will turn 19 years old during the trial for which there is no reference data above the age of 19 years (228 months). In these cases, the reference data for being 19 years old will be used.

## 2.5.3 IWQOL-Kids

The Impact of Weight on Quality of Life (IWQOL)-Kids questionnaire contains 27 questions (also referred to as items) with five response options ranging from never true (1) to always true (5). The 27 items are categorised into four scales: physical comfort (six items); body esteem (nine items); social life (six items); and family relations (six items).

The score on each scale will calculated as an unweighted sum of that scale's constituent items and then transformed to 0 to 100 scoring, where 100 represents the best quality of life, and 0 represents the worst quality of life. At least 50% of the items within a scale should be answered to calculate the scale score. For computation of the total score, the unweighted sum of all of the items will be used, and then scores will similarly transformed to the 0 to 100 scoring. At least 75% of the 27 items should be answered to calculate the total score.

| VV-TMF-4906149 | 1.1 | NN9536 | - | 4451 |
|----------------|-----|--------|---|------|
|----------------|-----|--------|---|------|

Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 Version: 1.0
Status: Final 

## 3 Changes to the statistical analyses planned in the protocol

The main analyses were described in the protocol for the trial NN9536-4451. However, clarifications and more detailed descriptions of endpoints and analyses are provided in this SAP. The changes from the protocol of NN9536-4451 are:

- Treatment-emergent hypoglycaemic episodes will also be classified according to ADA/ISPAD 2018<sup>4</sup> classification
- Fasting plasma glucose and lipids have been promoted from exploratory endpoints to supportive secondary endpoints in order to align with the upcoming STEP Young trial
- Based on feedback from authorities ALT has been promoted to a supportive secondary endpoint
- It is clarified that RD-MI imputation is performed with timing of last available observation during the on-treatment period (LAO-OT) added in the model as a covariate. This is true for all endpoints. This is to clarify that the grouping of subjects according to timing is as in McEvoy<sup>5</sup>
- It is clarified that TP-MI imputation is performed with penalties applied to both treatment arms
- Due to the stadiometer not being calibrated at site , a sensitivity analysis of the primary endpoint has been added
- A sensitivity analysis of the primary endpoint using an ANCOVA assuming unequal variances in the treatment arms has been added
- It is clarified that, in addition to OR, ETD will be reported for logistic regression analyses
- It is clarified that analyses of safety endpoints will be performed based on the safety analysis set
- It is specified that lipids, FPG and fasting insulin will also be analysed in SI-units
- Subgroup analyses of the primary and confirmatory secondary endpoint have been added due to a similar request from the authorities on the SCALE TEENS trial.

VV-TMF-4906149 | 1.1 | NN9536 - 4451

Statistical Analysis Plan
Study ID: NN9536-4451


Date: 16 December 2021 Version: 1.0
Status: Final 

## 4 References

- Centers for Disease Control and Prevention. Stature-for-age charts, 2 to 20 years, LMS
  parameters and selected smoothed stature percentiles in centimeters, by sex and age
  [Internet] 2018 [Cited August 2018].
- 2. World Health Organization. World Health Organization: Growth reference 5-19 years. Accessed at: <a href="http://www.who.int/growthref/who2007">http://www.who.int/growthref/who2007</a> bmi for age/en/ [updated 2 March 2018; cited 2018 2 March].
- 3. Ly TT, Maahs DM, Rewers A, Dunger D, Oduwole A, Jones TW, et al. ISPAD Clinical Practice Consensus Guidelines 2014. Assessment and management of hypoglycemia in children and adolescents with diabetes. Pediatr Diabetes. 2014;15 Suppl 20:180-92.
- Mayer-Davis EJ, Kahkoska AR, Jefferies C, Dabelea D, Balde N, Gong CX, et al. ISPAD Clinical Practice Consensus Guidelines 2018: Definition, epidemiology, and classification of diabetes in children and adolescents. Pediatr Diabetes. 2018;19 Suppl 27:7-19.
- 5. McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6.

24 of